CLINICAL TRIAL: NCT06804382
Title: Academic Detailing to Optimize PrEP Implementation in Pediatric Primary Care Settings: ADOPT-PrEP
Acronym: ADOPT-PrEP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Carly Guss, Assistant Professor, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB-P00050424
Record Dates: First submitted 2025-01-22; First posted 2025-02-03 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: PrEP; HIV Prevention Program
Keywords: PrEP; STI; AYA; adolescent; hiv prevention; academic detailing
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pediatricians (Experimental)
  Interventions: Behavioral: Academic detailing

INTERVENTIONS:
Behavioral: Academic detailing — Academic detailing is an evidence-based, 1-on-1 outreach education technique intended to promote clinician behavior change. Information gained during earlier focus groups will be used to develop study-specific materials.

SUMMARY:
In this study, 50 pediatricians will participate in academic detailing, an evidence-based, 1-on-1 outreach education technique intended to promote clinician behavior change through brief, highly interactive, and individualized dialogues with trained educators, or "detailers". The goals of this study are to learn about whether this is a practical and acceptable technique, and whether it changes how pediatricians prescribe pre-exposure prophylaxis (PrEP) to adolescents and young adults (AYA) and how patients take it.

DETAILED DESCRIPTION:
Adolescents and young adults (AYA) account for nearly 20% of new HIV diagnoses in the US. Only 10% of sexually active adolescents have ever been tested for HIV2 and very few have used pre-exposure prophylaxis (PrEP), despite it being safe, highly effective at preventing HIV transmission, and FDA-approved for youth. Pediatric health care providers (physicians and associate clinicians) could have a major impact on PrEP use for youth, as they are trusted sources of health information for AYA. However, pediatricians infrequently discuss or recommend PrEP due to limited training in sexual health and PrEP and a lack of tools and protocols to help them integrate PrEP into busy clinical workflows. Academic detailing, an evidence-based, 1-on-1 educational outreach technique for clinicians proven to change prescribing behaviors, could improve PrEP prescribing and persistence for AYA. Academic detailing has been associated with substantial increases in PrEP prescribing in adult settings but has not been tested in pediatric settings. The objective of this study is to develop an implementation strategy to improve PrEP provision to AYA at a large children's hospital and affiliated community health center in an HIV priority jurisdiction. Our hypothesis is that academic detailing for PrEP that has been adapted for a pediatric and young adult population will be feasible, acceptable, and result in rapid, sustained, and clinically significant improvements in PrEP provision in pediatric settings.

After conducting qualitative interviews with AYA and pediatric providers to explore barriers and facilitators and to them develop materials specific to this study, we will conduct a pilot study of academic detailing amongst 50 pediatric providers in the Boston area. Providers will be recruited from Boston-area practices and invited to participated in the pilot project. Providers will complete 2 academic detailing visits and a post-visit qualitative interview and survey to assess feasibility and acceptability. Secondary outcomes include preliminary impact of academic detailing on their knowledge, intentions and readiness to prescribe PrEP, and changes in PrEP prescriptions, persistence, and HIV testing after the intervention through electronic medical record review.

ELIGIBILITY:
Inclusion Criteria:

* Primary care provider at one of our 3 study sites (Boston Children's Hospital Adolescent/Young Adult Medicine, Martha Eliot Health Center, Children's Hospital Primary Care Center)

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2027-04-01 (Estimated); Primary Completion 2030-03-30 (Estimated); Study Completion 2030-03-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility | From enrollment to end of study interview at 4 months
  Feasibility will be assessed using survey question from other academic detailing campaigns and assessed on a 5-point Likert scale. Questions will be: "the key messages are feasible to implement in my practice" (1= not at all through 5= extremely)
Feasibility | From enrollment to end of second academic detailing session at 1 month
  Feasibility of academic detailing based on number of enrolled providers who complete both academic detailing visits
Acceptability | From enrollment to end of second academic detailing visit at 1 month.
  Acceptability of academic detailing as measured by provider satisfaction with the academic detailing visit. This will be assessed via the Prescriber Satisfaction with Academic Detailing questionnaire (PSAD). Answers are on a 5 point Likert scale (1=not at all through 5=extremely).
Acceptability | From enrollment to end of second academic detailing session at 1 month
  Acceptability of academic detailing based on completion of academic detailing sessions

SECONDARY OUTCOMES:
Impact of academic detailing on PrEP knowledge and prescribing | From enrollment to end of study interview at 4 months
  Preliminary impact of academic detailing on their knowledge, intentions and readiness to prescribe PrEP. This will be assessed via adapted questionnaires from other academic detailing campaigns. Questions will be assessed on a 5 point Likert scale (1=strongly agree through 5= strongly disagree). Example questions include: "I am or would be comfortable prescribing and managing patients on PrEP;" "I am willing to talk to my patients about PrEP if it might be indicated."
Change in PrEP Prescriptions | From 6 months prior to enrollment to 6 months after intervention
  Changes in PrEP prescriptions provided by participants to their patients by review of electronic medical record following academic detailing intervention. This will include refills of oral PrEP medications and on-time injections of injectable PrEP.
HIV Testing | From 6 months prior to enrollment to 6 months after academic detailing intervention
  Participant rates of HIV testing of their patients by review of the medical record.
Fidelity to intervention | From enrollment to end of second academic detailing visit at 1 month.
  Fidelity will be assessed by having academic detailers observe each other and then will provide feedback on adherence to academic detailing procedures by using a structured checklist (e.g., detailer delivers key messages, seeks commitment to behavior change from pediatrician).

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to participant privacy and data de-identification needs.

REFERENCES:
- [Background] Krakower DS, Naja-Riese GM, Edelstein ZR, Gandhi AD, Wahnich A, Fischer MA. Academic Detailing to Increase Prescribing of HIV Pre-exposure Prophylaxis. Am J Prev Med. 2021 Nov;61(5 Suppl 1):S87-S97. doi: 10.1016/j.amepre.2021.05.030. PMID 34686295